CLINICAL TRIAL: NCT03016091
Title: A Phase II, Open-label, Single Arm Trial of Pembrolizumab for Refractory Atypical and Anaplastic Meningioma
Brief Title: A Trial of Pembrolizumab for Refractory Atypical and Anaplastic Meningioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrural, dismal results
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-415
Record Dates: First submitted 2016-12-22; First posted 2017-01-10 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2018-01

CONDITIONS: Atypical Meningioma; Anaplastic Meningioma; Hemangiopericytoma
MeSH Terms: conditions — Meningioma; Hemangiopericytoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): IV Pembrolizumab 200mg, given every 3 weeks until disease progression or intolerable toxicity
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — anti PD-L1

SUMMARY:
A Phase II, Open-label, Single Arm Trial of Pembrolizumab for Refractory Atypical and Anaplastic Meningioma

DETAILED DESCRIPTION:
This is a multicenter, prospective, single arm, open label, interventional study. The goal of this study, is to evaluate feasibility and efficacy of pembrolizumab for the treatment of recurrent or progressive meningioma (WHO grades II-III) or hemangiopericytoma (HPC). All patients will receive IV pembrolizumab, at a dose of 200mg, every 3 weeks. Patients will be treated until disease progression or intolerable toxicity. Treatment can be stopped after one year of treatment in case of stable disease or completer response, with re-initiation of treatment upon progression. Expression of PD1 and PD-L1 will be tested, on tumor cells, using IHC staining on biopsy material obtained from previous surgeries.

All patients will have a baseline neurologic and clinical exam, MRI scan, a brain dedicated CT-PET scan, a baseline cognitive exam and QOL assessment with a dedicated questionnaire. Patients will have a clinical and neurological exam every treatment cycle. MRI scan will be repeated after 2 months from the beginning of the trial drug administration and then every 2-3 months. There are no designated and specific criteria for response assessment in the treatment of meningioma. Therefore, response evaluation will be made using the RECIST 1.1 criteria, as used for solid tumors. The trial will allow the continuation of pembrolizumab in case of stable or improved clinical response, when pseudo-progression is suspected in the MRI. In addition, response assessment will also be made according to the RANO criteria, as used for high grade glioma. This will be compared to the RECIST evaluation, but will not be used for treatment decision making.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Histologically, previously proven, grade II or III meningioma, HPC or classic radiographic features of a recurrent surgically inaccessible atypical or anaplastic meningioma.
5. All patients would have to have recurrence despite radiotherapy, unless radiotherapy is contraindicated.
6. No limit on the number of prior surgeries, radiation or radiosurgery treatments.
7. No limit on prior systemic therapies - chemotherapy or biological agents.
8. Patients who received stereotactic radiosurgery (SRS) are eligible without histologic documentation of recurrence if at least 6 months have passed from previous SRS treatment, and preferably, but not necessarily a 2-ﬂuoro-2-deoxy-D-glucose PET imaging demonstrated hypermetabolism.
9. KPS≥50%
10. At least 4 weeks since any prior therapy.
11. Life expectancy of at least 4 months.
12. Dexamethasone use will be allowed up to a dose of 2mg per day. Steroids dose should be reduced or stopped 7 days prior to treatment with study drug.
13. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

    Table 1 Adequate Organ Function Laboratory Values

    Hematological Absolute neutrophil count (ANC)≥1,500 /mcL Platelets≥100,000 / mcL Hemoglobin≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl)≤1.5 X upper limit of normal (ULN) OR

    ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

    ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

    Activated Partial Thromboplastin Time (aPTT)≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

    ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants a Creatinine clearance should be calculated per institutional standard.
14. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
15. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
16. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Patients who are steroid dependent and cannot reduce the dexamethasone dose to a maximal dose of 2mg per day.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 adult patients with histologically or radiologically proven recurrent or progressive meningioma (grade I to III) or anaplastic SFT who were treated in a single institution from 2018 to 2022 (15 patients with recurrent meningioma and 3 with anaplastic SFT). Patients were recruited at least 6 months after treatment with stereotactic radiosurgery.
Groups:
- Arm 1: IV Pembrolizumab 200mg, given every 3 weeks until disease progression, intolerable toxicity or up to 2 years of treatment.
  Pembrolizumab: anti PD-L1 18 patients received treatment
Period: Overall Study
Arm/Group | Arm 1
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 18
Age, Customized [Median (Full Range); unit: years] | 64.5 [28 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
KPS at baseline [Median (Full Range); unit: units on a scale] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. Maximum score is 100 - Normal; no complaints; no evidence of disease.
  Minimum score is 0 - Dead. More examples: 60-Requires occasional assistance but is able to care for most of their personal needs. 50 -Requires considerable assistance and frequent medical care.
  units on a scale | 60 [50 to 90]
Tumor type [Count of Participants; unit: Participants]
  Recurrent grade I meningioma | 3
  Atypical meningioma | 11
  Anaplastic meningioma | 1
  Anaplastic solitary fibrous tumor | 3
Multifocal disease [Count of Participants; unit: Participants] | 14
Number of previous surgeries [Median (Full Range); unit: surgeries] | 3 [2 to 7]
Number of previous radiation therapy courses [Median (Full Range); unit: radiation therapy courses] | 2 [1 to 3]
Number of previous systemic therapies [Number; unit: systemic therapies] | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: 6 months PFS refers to the percentage of patients in a study who remain alive and whose disease has not worsened 6 months after starting treatment.
  To determine the 6 months PFS rate for patients with recurrent or progressive meningioma on pembrolizumab therapy we used the RANO meningioma criteria. The Response Assessment in Neuro-Oncology meningioma criteria are guidelines used to evaluate treatment response in meningioma patients, incorporating both radiological and clinical factors. Tumor response is classified into categories such as: complete response (CR), where the tumor disappears. Partial response (PR) with a 50% or more reduction in tumor size. Minor response (MR) between 25% to 50% reduction in tumor size. Stable disease (SD) indicating minimal change, and progressive disease (PD) defined by at least a 25% increase in tumor size, new lesions, or worsening clinical symptoms. these criteria emphasize the use of consistent imaging techniques such as MRI.
Time Frame: 6 months after starting treatment
Population: all participants who were assigned to the group
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 18
Participants | 2

2. Primary Outcome: Progression Free Survival (PFS)
Description: 12 months PFS refers to the percentage of patients in a study who remain alive and whose disease has not worsened 12 months after starting treatment.
  To determine the 12 months PFS rate for patients with recurrent or progressive meningioma on pembrolizumab therapy we used the RANO meningioma criteria. The Response Assessment in Neuro-Oncology meningioma criteria are guidelines used to evaluate treatment response in meningioma patients, incorporating both radiological and clinical factors. Tumor response is classified into categories such as: complete response (CR), where the tumor disappears. Partial response (PR) with a 50% or more reduction in tumor size. Minor response (MR) between 25% to 50% reduction in tumor size. Stable disease (SD) indicating minimal change, and progressive disease (PD) defined by at least a 25% increase in tumor size, new lesions, or worsening clinical symptoms. these criteria emphasize the use of consistent imaging techniques such as MRI.
Time Frame: 12 months after starting treatment
Population: all participants who were assigned to the group
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 18
Participants | 2

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is a term used in reference to treatments for cancer. It refers to the time which begins at diagnosis and up to the time of death.
Time Frame: from date of diagnosis until date of death from any cause
Population: all participants who were assigned to the group
Measure: Median (Full Range); unit: month
Arm/Group | Arm 1
Number analyzed (Participants) | 18
month | 40 [2 to NA] — several patients were still alive at the end of the study

4. Secondary Outcome: Overall Progression Free Survival (PFS)
Description: To determine the overall progression free survival (PFS) rate for patients with recurrent or progressive meningioma on pembrolizumab therapy we used the RANO meningioma criteria. The Response Assessment in Neuro-Oncology meningioma criteria are guidelines used to evaluate treatment response in meningioma patients, incorporating both radiological and clinical factors. Tumor response is classified into categories such as: complete response (CR), where the tumor disappears. Partial response (PR) with a 50% or more reduction in tumor size. Minor response (MR) between 25% to 50% reduction in tumor size. Stable disease (SD) indicating minimal change, and progressive disease (PD) defined by at least a 25% increase in tumor size, new lesions, or worsening clinical symptoms. these criteria emphasize the use of consistent imaging techniques such as MRI.
Time Frame: From the initiation of treatment to the occurrence of disease progression or death.
Population: all participants who were assigned to the group
Measure: Median (Full Range); unit: month
Arm/Group | Arm 1
Number analyzed (Participants) | 18
month | 2.2 [1.9 to 27]

ADVERSE EVENTS:
Time Frame: Serious and other (Not Including Serious) Adverse Events were assessed from the beginning of treatment for up to two year, and all-cause mortality were assessed from the diagnosis until 1/12/2022.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 4/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=18)
Fatigue (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Twenty-five patients were required for the analysis to have 80% power to detect improvement in PFS-6 from 5% to 25% with a significance level of 0.05, and accounting for a 10% drop-out rate. The study was terminated after accrual of 18 patients, due to slow accrual and lack of efficacy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03016091/Prot_SAP_000.pdf